CLINICAL TRIAL: NCT02836899
Title: Prevention of Acute Kidney Injury by Nitric Oxide in Prolonged Cardiopulmonary Bypass. A Double Blind Controlled Randomized Trial in Cardiac Surgical Patients With Endothelial Dysfunction.
Brief Title: Effect of Nitric Oxide in Cardiac Surgery Patients With Endothelial Dysfunction.
Acronym: MGHK23
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ichinose, Fumito, M.D., Ph.D., Massachusetts General Hospital (Unknown); Kenneth, Shelton, M.D., Massachusetts General Hospital (Unknown); Kacmarek, Robert M., Ph.D., Massachusetts General Hospital (Unknown); Sundt, Thoralf M., M.D., Massachusetts General Hospital (Unknown); Villavicencio-Theoduloz, Mauricio A., M.D., Massachusetts General Hospital (Unknown); Thompson, Boyd Taylor, M.D., Massachusetts General Hospital (Unknown); Bonventre, Joseph V., M.D., Brigham Women Hospital (Unknown); Shann, Kenneth G., Massachusetts General Hospital (Unknown); Zapol, Warren M., M.D. (Individual); Marrazzo, Francesco, M.D., Massachusetts General Hospital (Unknown); Spina, Stefano, M.D., Massachusetts General Hospital (Unknown); Zadek, Francesco, M.D., Massachusetts General Hospital (Unknown); Rezoagli, Emanuele, M.D., Massachusetts General Hospital (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Lorenzo Berra, MD, Assistant Professor, Department of Anesthesia, Critical Care and Pain Medicine, Massachusetts General Hospital, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MGH K23; K23HL128882-01 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; nitric oxide; cardiopulmonary bypass; endothelial dysfunction; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Inhaled nitrogen will be administered via the cardiopulmonary bypass (CPB) machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the Intensive Care Unit (ICU). Once patients are extubated they will breathe test gas via a facemask or nasal cannula. Test gas administration will commence at the onset of CPB and last for 24 hours.
  Interventions: Other: Placebo
- Nitric Oxide (Experimental): Inhaled nitric oxide (iNO) will be administered via the CPB machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the ICU. Once patients are extubated they will breathe test gas via a facemask or nasal cannula. Test gas administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, iNO will be weaned and discontinued while carefully monitoring hemodynamics for a period of 2-4 hours.
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Inhaled nitric oxide will be administered in a final concentration of 80 ppm. The treatment will begin at the onset of the cardiopulmonary bypass until to 24h after Intensive Care Unit (ICU) admission, including 2-4 hours of weaning from nitric oxide and careful hemodynamics monitoring.
  Arms: Nitric Oxide
Other: Placebo — This is the placebo group. Nitrogen will be added instead of nitric oxide.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether nitric oxide is effective in the treatment of acute kidney injury in cardiac surgical patients with sign and laboratory data suggesting endothelial dysfunction undergoing prolonged cardiopulmonary bypass.

DETAILED DESCRIPTION:
I. SUBJECT ENROLLMENT

1. Methods of enrollment, including procedures for patient registration. Patients will be screened in the "Cardiac surgery pre-operative clinic", Massachusetts General Hospital (MGH) Cox building floor 6 (before surgery). If the patient is eligible and after obtaining the consent of the primary cardiac surgeon, the patient will be approached for consent to participate in this clinical trial. Consent will be obtained exclusively from the patient, and not from a surrogate, because cardiac surgery is usually a scheduled procedure. The obtaining of the consent directly from the patient is preferred, since there will be the opportunity of interaction with the patient when he/she is fully awake. After consent is obtained, the patient will be randomized to the study group. A de-identified code will be assigned to the patient and registered on a dedicated enrollment log.
2. Procedures for obtaining informed consent (including timing of consent process). Patients will be screened in the "Cardiac surgery pre-operative clinic", MGH Cox building floor 6 (before surgery). If a patient is eligible for the study and after obtaining the consent of the primary cardiac surgeon, the patient will be approached to consent to participate in the clinical trial. There is no need for surrogate consent for this trial, as explained above. Signing the Informed Consent Form will be requested for participation in the study. Personal Medical Information (PMI) will be accessed by the investigator(s) only for study purposes. Patients who choose not to participate in this study will receive standard care according to the procedures of the ICU, without any repercussion.
3. Treatment assignment and randomization (if applicable). To ensure a robust and unbiased approach, randomization should account for demographic characteristics of the patients (i.e.: age, sex) and glomerular filtration rate (GFR). Only patients who are cared for by experienced anesthesiologists and cardiac surgeons (more than 5 years of staff experience) will participate in this study. The patients will be randomized to receive either NO (study drug) or N2 (placebo) alone. In order to account for an elevated baseline pulmonary artery pressure, patients with pre-operative mean PAP ≥30 mmHg will be allocated equally to the two groups during the stratified randomization process. The random allocation sequence will be created using a computerized random generation program. The randomization will be in blocks of 10 patients. The intervention will consist of administering the test gas via the cardiopulmonary bypass (CPB) machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the Intensive Care Unit (ICU). When patients are extubated they will breathe test gas via a facemask or nasal prongs. Test gas administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, inhaled NO (iNO) will be weaned and discontinued while carefully monitoring hemodynamics for a period of 2-4 hours. Local guidelines for NO gas discontinuation will be followed. Using commercially available tanks of Nitric Oxide (Airgas Inc, Radnor Township, Pennsylvania) or volumetrically-calibrated flowmeters, pure N2 (placebo) or 850 ppm NO gas in N2 will be mixed with pure oxygen (O2) or air to obtain the desired concentration of O2 and, in the NO treatment group, a final concentration of 80 ppm NO. For safety, nitric oxide, nitrogen dioxide (NO2), O2 and methemoglobin (Met-Hb) levels will be continuously monitored by the personnel unblinded to the study. Patients in the placebo (N2) group will receive nitrogen test gas during the same 24 hour-period. The inspired oxygen levels will be maintained at the usual levels required for routine post-operative care. No changes to the usual and customary standards of care for any intraoperative or postoperative treatment will be made during the study period.
4. Blinding procedure for Nitric Oxide and Nitrogen delivery. A double-blind study will be performed to avoid potential patient and investigator bias, the study is blinded to: participants, perfusionists, surgeons, anesthesiologists, ICU physicians and the nursing staff. The test gas tank and the gas delivery system in the operating room (OR) and at the bedside will be masked. The respiratory therapist in the ICU and a member of the study staff will be unblinded and will prepare the appropriate test gas tanks and NO/N2 meters. Blood Met-Hb levels and NO/NO2 concentrations are safety concerns that the respiratory therapist and one member of the study staff will monitor and regulate (NO2 levels will be maintained below 5 ppm, and Met-Hb below 5%, if necessary by reducing NO concentration to 40 ppm or less according to MGH guidelines NO therapy).

II. STUDY PROCEDURES a. Study visits and parameters to be measured (e.g., laboratory tests, x-rays, and other testing). SCREENING visit: Screening will take place in the "Cardiac surgery pre-operative clinic", MGH Cox building floor 6 (before surgery). Patients will be screened if they require prolonged CPB (>90 minutes on CPB, i.e., valve replacement ± coronary artery bypass grafting (CABG)) and if the primary cardiac surgeon of the patient agrees on enrolling the patient in the study.

Screening consists of:

* Review eligibility entry criteria of the study: inclusion/exclusion criteria will be reviewed.
* Review the research protocol: This is a protected time for the subject to ask questions and become familiar with all aspects of the study protocol.
* Administration of a brief questionnaire to determine endothelial function with the subject verbal assent on the day of pre-surgical evaluation. The questionnaire evaluates medical history, integrating clinical and laboratory data of screened patients. In males > 40 year old and females > 50 year old, endothelial dysfunction has been shown to be associated with at least one the following criteria: Previous coronary artery bypass graft or PTCA (+ stent); History or presence of intermittent claudication; Critical limb ischemia, or peripheral vascular disease with the Exception of vasculitis; History of transient ischemic attack and/or ischemic stroke; Diagnosis of diabetes (IDDM or NIDDM) requiring oral hypoglycemic agents or insulin; Hypercholesterolemia (total cholesterol > 200 mg/dl or LDL > 160 mg/dl) treated with statins, ion- exchange resins or other oral agents; BMI > 40; Hypertension (SBP 140 ≥ mmHg) treated with antihypertensive drugs; Active smoking ≥ 10 pack - years
* Consent form: The subject will be asked to sign the consent form.

Laboratory tests will be reviewed by the same physician, and if inclusion/exclusion criteria are met, subjects will be enrolled.

RANDOMIZATION. Patients will be randomly allocated to one of the test gas study groups (inhaled 80 parts per million (ppm) nitric oxide in nitrogen) or the placebo group (inhaled N2). The intervention will consist of giving the test gas both via the CPB machine and after CPB via the anesthetic circuit, and thereafter via the mechanical ventilator and/or with face mask/nasal prongs in the ICU/ward. Test gas administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, iNO will be weaned and discontinued while carefully monitoring hemodynamics for a period of 2-4 hours. Local guidelines for iNO discontinuation will be adopted. Using an Inovent (Ikaria Inc, N.J., USA) or volumetrically-calibrated flowmeters, pure nitrogen (placebo) or 850 ppm NO gas in N2 is mixed with pure O2 or air to obtain a final concentration of 80 ppm NO. During CPB the test gas is delivered through the extracorporeal oxygenator, after CPB the NO is delivered through the inspiratory limb of the anesthetic or ventilator circuit. NO, NO2 and O2 and methemoglobin levels are monitored by an unblinded observer. Patients in the placebo group will receive nitrogen test gas during the same 24 hour-period. When patients are extubated they will breathe test gas via a face mask or nasal prongs. The inspired oxygen levels will be maintained at the usual levels required for routine post-operative care. The test gas tank in the OR and at the bedside will be covered and blinded from the clinicians treating the patient. Only the respiratory therapist in the ICU and a member of the study staff will be unblinded and will prepare the appropriate test gas tanks and NO/N2 meters. No changes to the usual and customary standards of care for any intraoperative or postoperative treatments will be made during the study period.

III. MONITORING AND QUALITY ASSURANCE

1. Independent monitoring of source data. Informed consent forms, case report forms, and data will be reviewed by the principal investigator following enrollment of every 5 subjects and an independent data and safety monitor following enrollment of every 50 subjects to the protocol to ensure safety of the study subjects. The safety data that will be reviewed includes: patient-, nurse-, research-assistant, or investigator-reported adverse events such as reason for early termination of the protocol, or adverse reaction to NO. Other data to be reviewed includes appropriate handling and processing of blood samples and maintenance of patient confidentiality throughout the study.
2. Safety monitoring (e.g., Data Safety Monitoring Board, etc.). An interim analysis by a Data Safety management Board (DSMB) comprised of 3 members is planned at reaching 50% of the study population (125 patients enrolled). The study will only be stopped if the interim analysis detects a significant increase of mortality, acute kidney injury (AKI), need for renal replacement therapy (RRT), myocardial infarction (MI), post-operative hemorrhage, other significant morbidity in the NO test gas group.

   Members of the Data Safety Management Board (DSMB) consist of an anesthesiologist with clinical expertise in NO, a cardiologist and a nephrologist.
3. Outcomes monitoring. Plasma creatinine will be measured daily until day 7 after CPB or until discharge from the hospital if this occurs earlier. Urine output will be assessed until day 7 after CPB or until discharge from the hospital if this occurs earlier. Follow up will be completed at 1 year after surgery as described in "V. Study procedure".
4. Adverse event reporting guidelines. The principal investigator will review any adverse events immediately following their occurrence and report them to the Institutional Review Board (IRB) in accordance with Partners Investigator guidelines. Specifically, for this study, serious adverse events will be reported by phone, fax, or email within 24 hours to the Human Research Committee (HRC), followed by a full written report within 10 business/14 calendar days. Mild or moderate adverse events will be presented in progress reports at continuing reviews.

Stopping rules. The review and decision regarding altering or stopping the protocol will be performed by the principal investigator together with the DSMB. Mild or moderate adverse events will be presented in progress reports at continuing reviews. Protocol exit criteria will be:

1. Acute worsening hypotension: decrease in mean blood pressure of > 20 mmHg not attributable to other causes, i.e., hypovolemia, hemorrhage, sepsis, acute heart failure.
2. Sudden worsening of hypoxemia: decrease of peripheral oxygen saturation (SatO2) < 70% at 100% of inspiratory oxygen fraction (FiO2) not attributable to other causes, i.e., pulmonary edema, acute respiratory distress syndrome (ARDS), pulmonary embolism.
3. An increase in NO2 levels > 5 ppm from baseline or any life-threatening symptom potentially attributed to NO administration by the physician investigator.

IV. BIOSTATISTICAL ANALYSIS

a. Specific data variables being collected for the study

Preoperative collection of patient data from the MGH electronic medical chart (EPIC) will include:

* Patient demographics
* Past and current medical and surgery history and therapy
* Co-morbidities
* Pertinent cardiopulmonary test results: i.e., echocardiography, cardiac catheterization, pulmonary function tests, and chest imaging).

Prospective collection of patient data will include:

* ICU and length of hospital stay
* Duration of mechanical ventilation
* Hospital course
* Intrahospital mortality and mortality at 6 weeks, 90 days and 1 year after cardiac surgery.
* Activity of daily living at and postoperative health related quality of life (PROMIS questionnaire for global health) at 6 weeks, 90 days and 1 year after surgery.
* Nonfatal stroke before surgery and at 6 weeks after surgery
* Perioperative and non-perioperative nonfatal myocardial infarction, as defined by the third universal definition of MI released in 2012 by the European Society of Cardiology (ESC)/American College of Cardiology Foundation (ACCF)/American Heart Association (AHA)/World Heart Federation (WHF)
* Renal failure requiring dialysis at any time during hospitalization and at 6 weeks, 90 days and 1 year after cardiac surgery.
* Acute Kidney Injury as difened by KDIGO criteria.
* Organ dysfunction assessed daily in ICU by using Sequential organ failure assessment (SOFA).
* Delirium assessed daily in the first 7 days after surgery by using the confusion assessment method for intensive care unit (CAM-ICU).
* Cardiovascular support: vasopressors and inotropic agents requirement (Vasoactive-inotropic score), need for balloon pump or ventricular-assist device.
* Post-operative infections, cardiac arrhytmias and non cardiac complications.

Samples to be collected:

1. Blood samples will be collected before surgery, at the end of surgery, each day until day 7 after the cardiac procedure or until hospital discharge if before day 7, and at 6 weeks. The samples will be tested for: creatinine (after surgery, 24 hours after the end of CPB, 48 hours after the end of CPB, POD3, POD4, POD5, POD6, POD7 and 6 weeks) and biomarkers for kidney injury (immediately before CPB, 15 minutes after the end of CPB, 24 hours after the end of CPB, 48 hours after the end of CPB and at 6 weeks). Urine samples will be collected for urinary biomarkers of kidney injury immediately before CPB, 15 minutes after the end of CPB, 24 hours after the end of CPB, 48 hours after the end of CPB and at 6 weeks.
2. Statistical methods. The primary aim of this study is to determine whether supplementation with NO decreases the incidence of AKI in patients with signs and symptoms suggesting endothelial dysfunction. A total of 250 cardiac-surgery patients will be enrolled, requiring more than 90 minutes of CPB. The two arms will be compared for homogeneity of baseline characteristics (age, weight, sex, and GFR), intraoperative course (CPB time, amount of blood transfusions) and postoperative data (post-operative transfusions, adverse events directly related to surgery procedures). To examine differences between the two groups, we will use an unpaired Student's t-test for continuous variables with a normal distribution, a Mann-Whitney U test for continuous variables that are not normally distributed and a Fisher's exact test for dichotomous variables. Continuous variables will be described as mean±standard deviation (SD) when normally distributed, median with interquartiles (IQR) when not normally distributed, or count (%) if a dichotomous variable. The change in the laboratory markers over time and between the two groups will be tested with a repeated measures ANOVA. The incidence of AKI and postoperative adverse events after prolonged CPB will be described in terms of relative risk with significance level and confidence intervals for the two groups. Based on the occurrence of missing data, the strategy to manage them will be decided. However, our aim would be not to use any kind of imputation.
3. Power analysis. The sample size of this trial was calculated based on the primary endpoint: the reduction of AKI incidence. Despite we do not have track incidence, AKI is very common in our MGH patients after open-heart surgery, and it is reasonable to assume that AKI incidence is similar to those recent reports from US and European studies at major academic centers CPB (AKI incidence has been reported to be between 50 to 60%). In our prior trial on NO in cardiac surgery, the sample size was calculated to find a 30% reduction in the incidence of AKI (n=212 in that trial). We estimate a greater (35%) reduction in the incidence of AKI because we anticipate that this population with signs and symptoms of endothelial dysfunction will be more affected by the beneficial therapeutic properties of NO. Thus, in the NO group the incidence of AKI is expected to decrease from 55% to 35.75%. The sample size needed to detect a difference, assuming an alpha error of 0.05 (two-sided test) and a study power of 0.8, is 114 patients per group. In order to account for possible dropouts, we increased our sample size by 10%. We will enroll 250 patients, 125 in the NO group and 125 patients in the control (N2) group.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Age ≥ 18 years of age
3. Elective cardiac or aortic surgery with CPB>90 minutes
4. Stable pre-operative renal function without evidence of plasma creatinine level increase of ≥ 0.3 mg/dL over the prior 3 months and without renal replacement therapy (RRT).
5. Clinical evidence of endothelial dysfunction assessed by a specifically designed questionnaire.

Exclusion Criteria:

1. eGFR less than 30 ml/min/1.73 m2
2. Emergent cardiac surgery.
3. Life expectancy < 1 year at the time of enrollment.
4. Hemodynamic instability as defined by a systolic blood pressure <90 mmHg.
5. Mean pulmonary artery pressure ≥ 40 mm Hg and PVR > 4 Wood Units.
6. Left ventricular ejection fraction < 30% by echocardiography obtained within three months of enrollment
7. Administration of one or more Packed Red Blood Cells (RBCs) transfusion in the week prior to enrollment.
8. X-ray contrast infusion less than 48 hours before surgery.
9. Evidence of intravascular or extravascular hemolysis from any other origin:

   i. Intravascular: Intrinsic RBCs defects leading to hemolytic anemia (eg, enzyme deficiencies, hemoglobinopathies, membrane defects). Extrinsic: liver disease, hypersplenism, infections (eg, bartonella, babesia, malaria), treatment with oxidizing exogenous agents (eg, dapsone, nitrites, aniline dyes), exposure to other hemolytic agents (eg, lead, snake and spider bites), lymphocyte leukemia, autoimmune hemolytic disorders.

   ii. Extravascular: Infection (eg, clostridial sepsis, severe malaria), paroxysmal cold hemoglobinuria, cold agglutinin disease, paroxysmal nocturnal hemoglobinuria, iv infusion of Rho(D) immune globulin, iv infusion of hypotonic solutions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | 7 days
  Incidence of Acute Kidney injury according to KDIGO criteria.

SECONDARY OUTCOMES:
AKI severity | 7 days after cardiac surgery
  Difference in AKI severity between the two groups using following KDIGO stages.
Renal replacement therapy | up to 1 year
  To study the incidence of acute renal failure requiring RRT
Major Adverse Kidney Events (MAKE) | 6 weeks after cardiac surgery
  Difference between groups of MAKE at 6 weeks after surgery. MAKE is a composite outcome of death, new dialysis and worsened renal function (defined as a 25% or greater decline in eGFR compared to the baseline).
Organ dysfunction | 7 days
  Assessment of organ dysfunction through the evaluation of SOFA score
Prolonged cardiovascular support | 48 hours after cardiac surgery
  Difference between groups of prolonged cardiovascular support defined as need for vasopressors, inotropic agents, balloon pump, or ventricular-assist device for more than 48 hours after cardiac surgery.
Vasoactive-inotropic score (VIS) | 7 days after cardiac surgery
  Difference between groups of maximum daily VIS and duration of vasopressors and or inotropic agents support. VIS is calculated as Dopamine dose (mcg/kg/min) + Dobutamine dose (mcg/kg/min) + 100 x Epinephrine dose (mcg/kg/min) + 10 x Milrinone dose (mcg/kg/min) + 10,000 x Vasopressin dose (units/kg/min) + 100 x Norepinephrine dose (mcg/kg/min) + 10 x Phenilephrine dose (mcg/kg/min).
Duration of mechanical ventilation | up to 6 weeks
  Difference of duration of mechanical ventilation
Intensive care unit length of stay (ICU-LOS) | up to 6 weeks
  Difference between groups of ICU-LOS defined as number of days spent in an ICU bed.
Hospital length of stay (LOS) | up to 1 year
  Difference between groups of hospital LOS defined as number of days spent in a hospital bed.

OTHER OUTCOMES:
Renal tubular injury | Up to 6 weeks
  Renal biomarkers to evaluate renal tubular injury.
Incidence of AKI related to risk factors | 7 days
  Incidence and severity of AKI related to presence of CKD at baseline, duration of CPB, duration of aortic cross clamp, levels of free Hb, levels of NO consumption, pulmonary pressure at baseline, cardiovascular risks associated with endothelial dysfunction, scheduled procedure and EuroSCORE II.
Incidence of delirium | 7 days after cardiac surgery
  Difference between groups of Incidence of Delirium will be assessed daily in the first 7 days after surgery by using the confusion assessment method for intensive care unit (CAM-ICU).
Score of the Activity of Daily Living | One year follow up
  Analysis of the quality of life up to 1 year after surgery by the Activity of Daily Living evaluation (by Katz Index) and PROMIS global health.
Overall mortality | up to 1 year
  Evaluation of the overall intrahospital mortality and at 28 6 weeks 90 days and 1 year after surgery
Methemoglobin levels in blood | During and 48 hours after cardiac surgery
  Blood methemoglobin levels will be measured to evaluate the oxidation of oxyhemoglobin in the two groups until 48h after surgery.
Incidence of non fatal stroke | 6 weeks
  Difference between groups of incidence of non fatal stroke will be assessed by at 6 weeks after cardiac surgery.
Perioperative and non-perioperative nonfatal myocardial infarction | 72 hours and 1 year follow up
  Incidence of Perioperative and non-perioperative nonfatal myocardial infarction as defined by the third universal definition of MI released in 2012 by the ESC/ACCF/AHA/WHF.
Post operative bleeding | 24 after surgery
  Incidence of postoperative bleeding calculated as the sum of blood loss through thoracic drains from the moment of closure of the chest over a period of 24 hours.
Transfusions | 7 days surgery
  Differences between the two groups of transfusions with plasma and stored or autologous red blood cells (RBCs) recovered using intraoperative cell salvage devices.
Post-operative infections | 6 weeks
  Post-operative infections (e.g., pneumonia, wound infection, endocarditis, central line infection, urinary tract infection, sepsis).
Cardiac and non-cardiac complications | 6 weeks
  Cardiac arrhythmias and other non-cardiac post-operative complications (e.g., hepatobiliary disorders, pneumothorax, pleural effusion, vascular disorders).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arora P, Di Fenza R, Shetty NS, Giammatteo V, Marrazzo F, Spina S, Zadek F, Gianni S, Fakhr BS, La Vita C, Shann K, Zheng H, Gaonkar M, Yu B, Feelisch M, Thompson TB, Akeju O, Sundt TM, Bonventre J, Ichinose F, Berra L; Cardiac Anesthesia Research Group. Nitric Oxide to Reduce Acute Kidney Injury in Patients with Pre-existing Endothelial Dysfunction Requiring Prolonged Cardiopulmonary Bypass: A Randomized Clinical Trial. Anesthesiology. 2025 Nov 21. doi: 10.1097/ALN.0000000000005861. Online ahead of print. PMID 41270263
- [Derived] Marrazzo F, Spina S, Zadek F, Lama T, Xu C, Larson G, Rezoagli E, Malhotra R, Zheng H, Bittner EA, Shelton K, Melnitchouk S, Roy N, Sundt TM, Riley WD, Williams P, Fisher D, Kacmarek RM, Thompson TB, Bonventre J, Zapol W, Ichinose F, Berra L. Protocol of a randomised controlled trial in cardiac surgical patients with endothelial dysfunction aimed to prevent postoperative acute kidney injury by administering nitric oxide gas. BMJ Open. 2019 Jul 4;9(7):e026848. doi: 10.1136/bmjopen-2018-026848. PMID 31278097
- See also: This is the clinical trial that we previously performed in collaboration with Xijing Hospital. — https://clinicaltrials.gov/ct2/show/study/NCT01802619?term=lize+xiong&rank=7